CLINICAL TRIAL: NCT02942264
Title: Phase I Trial of Zotiraciclib (TG02) Plus Dose-Dense or Metronomic Temozolomide Followed by Randomized Phase II Trial of Zotiraciclib (TG02) Plus Temozolomide Versus Temozolomide Alone in Adults With Recurrent Anaplastic Astrocytoma and Glioblastoma
Brief Title: Zotiraciclib (TG02) Plus Dose-Dense or Metronomic Temozolomide Followed by Randomized Phase II Trial of Zotiraciclib (TG02) Plus Temozolomide Versus Temozolomide Alone in Adults With Recurrent Anaplastic Astrocytoma and Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jing Wu, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 170009; 17-C-0009
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Brain Tumor; Astrocytoma; Astroglioma; Glioblastoma; Gliosarcoma
Keywords: Brain Tumor; Glioblastoma; Relapse; Randomized; Temodar
MeSH Terms: conditions — Brain Neoplasms; Astrocytoma; Glioblastoma; Gliosarcoma; Recurrence | interventions — 14-methyl-20-oxa-5,7,14,26-tetraazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8(27),9,11,16,21,23-decaene; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I Arm 1 Dose Dense Temozolomide plus Zotiraciclib (TG02) (Experimental): dose dense (dd) Temozolomide (TMZ) 125 mg/m^2 x 7 days on / 7 days off plus Zotiraciclib (TG02) dose escalation
  Interventions: Drug: Zotiraciclib (TG02); Drug: Temozolomide (TMZ)
- Phase I Arm 2 Metronomic Temozolomide Plus Zotiraciclib (TG02) (Experimental): metronomic Temozolomide (TMZ) 50 mg/ m^2 daily plus Zotiraciclib (TG02) dose escalation
  Interventions: Drug: Zotiraciclib (TG02); Drug: Temozolomide (TMZ)
- Phase II Arm 1 Maximum Tolerated Dose (MTD) of Zotiraciclib (TG02) Plus Temozolomide (TMZ) (Experimental): Maximum tolerated dose (MTD) of Zotiraciclib (TG02) from phase I plus and "winner" of dose dense (dd) vs metronomic Temozolomide (TMZ) from phase I
  Interventions: Drug: Zotiraciclib (TG02); Drug: Temozolomide (TMZ)
- Phase II Arm 2 Metronomic Temozolomide (TMZ) (Active Comparator): "winner" of dose dense (dd) vs metronomic Temozolomide (TMZ) from phase I alone
  Interventions: Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: Zotiraciclib (TG02) — Phase I: Two treatment arms and several dose levels are planned; In the maximum tolerated dose (MTD) finding part, Temozolomide (TMZ) with two alternate schedules (dose dense (dd) and metronomic (mn) in combination with Zotiraciclib (TG02) will be administered;
  --A cohort extension of both arms will be performed at each MTD and the treatment arm with a better progression free survival at 4 months (PFS4) will be selected for the combination treatment arm for Phase II; Patients will be randomized between two competing treatment arms: (winner of dd vs mn) TMZ + Zotiraciclib (TG02) versus dd/mn TMZ alone using a Bayesian clinical trial design. The dosage for the combination arm will be derived from the MTD determined in the Phase I component of the study.
  Other Names: TG02
  Arms: Phase I Arm 1 Dose Dense Temozolomide plus Zotiraciclib (TG02); Phase I Arm 2 Metronomic Temozolomide Plus Zotiraciclib (TG02); Phase II Arm 1 Maximum Tolerated Dose (MTD) of Zotiraciclib (TG02) Plus Temozolomide (TMZ)
Drug: Temozolomide (TMZ) — Phase I: In the maximum tolerated dose (MTD) finding part, Temozolomide (TMZ) with two alternate schedules (dose dense (dd) and metronomic (mn) in combination with Zotiraciclib (TG02) will be administered; A cohort extension of both arms will be performed at each MTD and the treatment arm with a better progression free survival at 4 months (PFS4) will be selected for the combination treatment arm for Phase II; Patients will be randomized between two competing treatment arms: ("winner" of dd vs mn) TMZ + Zotiraciclib (TG02) versus dd/mn TMZ alone using a Bayesian clinical trial design.
  Other Names: Temodar

SUMMARY:
Background:

Zotiraciclib (TG02) is an investigational drug that penetrates the blood-brain barrier and might treat brain tumors. Temozolomide (TMZ) is a drug used to treat brain tumors.

Objective:

To find out if Zotiraciclib (TG02) is safe, and to find out if it in combination with TMZ is as effective as TMZ alone in people with brain tumors.

Eligibility:

People ages 18 and older with a brain tumor that has progressed after standard treatment

Design:

In phase I part, the Bayesian optimal interval (BOIN) design will be used to find the maximum tolerated dose (MTD) of Zotiraciclib (TG02) for Arm 1 (dose dense TMZ) and Arm 2 (metronomic TMZ) independently. Then a randomized cohort expansion compared progression free survival at 4 months (PFS4) of the two arms for an efficient determination of a TMZ schedule to combine with Zotiraciclib at MTD.

In Phase II part, a Bayesian design based on posterior probability will be used to monitor efficacy.

Participants will be screened with:

* Medical history
* Physical exam
* Blood and urine tests
* Magnetic resonance imaging (MRI) of the brain if they have not had one in 14 days
* Heart test
* Tissue sample from prior surgeries

Participants will take Zotiraciclib (TG02) plus TMZ by mouth in 28-day cycles.

* Some will take TMZ for 7 days on and 7 days off. Others will take it every day.
* They will all take Zotiraciclib (TG02) three days before Cycle 1, and then on four days during every cycle.
* They will all get treatment to prevent vomiting and diarrhea before and for 24 hours after each Zotiraciclib (TG02) dose.
* They will all keep a diary of when they take the drugs and their symptoms.

Participants will have study visits. These include:

* Physical exam, heart test, quality of life questionnaire, brain MRI, and urine tests every 4 weeks
* Blood tests every 2 weeks

Participants will continue treatment until their disease gets worse or they have intolerable side effects.

Participants will also be enrolled in another protocol to test molecular markers for their brain tumor.

DETAILED DESCRIPTION:
Background:

* Zotiraciclib (TG02) is a pyrimidine-based multi-kinase inhibitor that has been shown to have inhibitory effects on cyclin-dependent kinases (CDKs), Janus Kinase 2 (JAK2) and Fm-like tyrosine kinase 3 (Flt3). It is orally administered and penetrates blood brain barrier (BBB). There is clinical experience in using Zotiraciclib (TG02) as both a single agent and in combination with other chemotherapy agents for cancer treatment.
* Temozolomide (TMZ) is an oral alkylating agent that has proven efficacy in anaplastic glioma and glioblastoma. It was approved by the United States (U.S.) Food and Drug Administration (FDA) to treat anaplastic astrocytoma and glioblastoma in adults. Both a dose-dense (dd) schedule, 7 days on and 7 days off and a metronomic (mn) daily dosing schedule have been used to treat recurrent high-grade gliomas.
* Our preclinical data have demonstrated that Zotiraciclib (TG02) down-regulates cyclin-dependent kinase 9 (CDK9) activity and its target proteins, such as anti-apoptotic protein myeloid-cell leukemia (Mcl-1), X-linked inhibitor of apoptosis (XIAP) and survivin. A treatment with Zotiraciclib (TG02) and TMZ has synergistic anti-glioma effects in a variety of glioma models with different genetic background. This serves as the basis for this proposed clinical trial.

Objectives:

Phase I:

-To determine the maximum tolerated dose (MTD) of Zotiraciclib (TG02) plus TMZ using both the dd and mn TMZ schedules in adult patients with recurrent anaplastic astrocytoma or glioblastoma/gliosarcoma.

To select the treatment regimen with better progression free survival (PFS)4 between Zotiraciclib (TG02) plus dd TMZ or mn TMZ at each of the MTDs following cohort expansion.

Phase II:

-To determine the efficacy of Zotiraciclib (TG02) plus TMZ versus TMZ alone in patients with recurrent World Health Organization (WHO) grade III or IV astrocytoma as determined by progression free survival.

Eligibility:

* Documented pathology diagnosis of anaplastic astrocytoma [WHO grade III], or glioblastoma/gliosarcoma (WHO grade IV) with recurrent disease. If the pathology diagnosis is anaplastic glioma or anaplastic oligoastrocytoma, evidence of either intact 1p/19q chromosomes or molecular features suggesting astrocytic tumor must be present. (including, but not limited to α-thalassemia mental retardation X-linked (ATRX) and/or tumor protein P53 (TP53) mutation)
* No prior use of bevacizumab as a treatment for brain tumor.
* No more than two prior relapses for Phase I and no more than one prior relapse for Phase II.
* Patients must have recurrent disease, either histologically proven or with imaging suggestive of recurrent disease
* Tumor tissues available for review to confirm the histologic diagnosis.
* Tumor tissue blocks available for molecular profiling analysis.

Design:

* Phase I:

  * This portion of the study is conducted in two stages: The MTD finding and cohort extension. Two treatment arms and several dose levels are planned.
  * In the MTD finding part, TMZ with two alternate schedules (dd and mn) in combination with Zotiraciclib (TG02) will be administered.
  * A cohort extension of both arms will be performed at each MTD and the treatment arm with a better progression free survival at 4 months (PFS4) will be selected for the combination treatment arm for Phase II.
  * Pharmacokinetic, pharmacogenetic studies and neutrophil analysis will be performed during the cohort extension of both arms.
  * A maximum of 72 patients will be enrolled to this component for the trial.
* Phase II:

  --Patients will be randomized between two competing treatment arms: ("winner" of dd vs mn) TMZ + Zotiraciclib (TG02) versus dd/mn TMZ alone using a Bayesian clinical trial design. The dosage for the combination arm will be derived from the MTD determined in the Phase I component of the study.
* The treatment schedule will be identical to that described above in the phase I component, with each cycle comprising 28 days.
* Patients will continue treatment until tumor progression or unacceptable toxicity occurs.
* At progression, patients randomized to the control arm (Temozolomide [TMZ] alone) will be offered the opportunity to continue TMZ and additional treatment with Zotiraciclib (TG02).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Inclusion criteria are same in both Phase I and Phase II parts, except for the number of prior disease relapses
* Patients must have pathologic diagnosis of anaplastic astrocytoma defined as World Health Organization (WHO) grade III or glioblastoma/gliosarcoma, WHO grade IV, which are confirmed by National Cancer Institute (NCI) Laboratory of Pathology. If the pathology diagnosis is anaplastic glioma or anaplastic oligoastrocytoma, evidence of either intact combined loss of the short arm chromosome 1 (i.e. 1p) and the long arm of chromosome 19 (1p/19q) chromosomes or molecular features suggesting astrocytic tumor must be present (including, but not limited to alpha-thalassemia/mental retardation, alpha-thalassemia/mental retardation, X-linked (ATRX), tumor protein P53 (TP53).
* Patients must have recurrent disease, histologically proven or imaging suggestive of recurrent disease as determined by principal investigator (PI). Prior implantation of Gliadel wafers is acceptable, if tumor recurrence is confirmed by histologic examination of the recurrent tumor
* Patients must have the ability to understand and the willingness to sign a written informed consent document.
* Patients must be greater than or equal to 18 years old.
* No more than two prior disease relapses to be eligible for the phase I portion of the study and no more than one prior relapse to be eligible for phase II.
* Patients must have undergone prior standard therapy for their primary disease. For patients with glioblastoma, this would include surgical resection, or biopsy, if safe resection was not permitted due to the tumor location, radiation and adjuvant temozolomide. For patients with anaplastic astrocytoma, this would include surgical resection, radiation and adjuvant chemotherapy procarbazine, lomustine (CCNU) and vincristine (PCV) or temozolomide.
* Tumor tissue must be available for review to confirm histological diagnosis.
* Tumor block or unstained slides must be available for molecular profiling.
* Karnofsky > 60 percent
* Patients must have adequate bone marrow function (absolute neutrophil count (ANC) > 1,500/mm^3, platelet count of > 100,000/mm^3), adequate liver function (alanine aminotransferase (ALT) and aspartate aminotransferase (AST)< 3 times upper limit normal and alkaline phosphatase < 2 times upper limit normal, total bilirubin < 1.5mg/dl), and adequate renal function (blood urea nitrogen (BUN) < 1.5 times institutional normal and serum creatinine < 1.5 mg/dl) prior to registration. These tests must be performed within 14 days prior to registration. Total bilirubin: patients with Gilbert's Syndrome are eligible for the study. (Total bilirubin level can be exempted from the eligibility criterion.)
* Patients must have recovered from the toxic effects of prior therapy to less than grade 2 toxicity per Common Terminology Criteria (CTC) version 4 (except deep vein thrombosis)
* At the time of registration, subject must be removed from prior therapy as follows:

  * greater than or equal to (28 days) from any investigational agent,
  * greater than or equal to 4 weeks (28 days) from prior cytotoxic therapy,
  * greater than or equal to 2 weeks (14 days) from vincristine,
  * greater than or equal to 6 weeks (42 days) from nitrosoureas,
  * greater than or equal to 3 weeks (21 days) from procarbazine administration,
  * greater than or equal to 1 week (7 days) for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. radiosensitizer does not count.
* Patients having undergone recent resection of recurrent or progressive tumor will be eligible given all of the following conditions apply:

  * At least 2 weeks (14 days) have elapsed from the date of surgery and the patients have recovered from the effects of surgery.
  * Evaluable or measureable disease following resection of recurrent malignant glioma is not mandated for eligibility into the study.
  * To best assess the extent of residual disease post-operatively, an magnetic resonance imaging (MRI) should be done no later than 96 hours in the immediate post-operative period or at least within 4 weeks post- operatively, within 14 days prior to registration. If the 96-hour scan is more than 14 days before registration, the scan needs to be repeated. The patient must have been on a stable steroid dose for at least 5 days prior to the baseline MRI. Steroids may be initiated as clinically indicated once baseline imaging has been completed with a goal of titrating steroids as soon as clinically warranted.
* Patients must have received prior radiation therapy and must have an interval of greater than or equal to 12 weeks (84 days) from the completion of radiation therapy to study entry except if there is unequivocal evidence for tumor recurrence (such as histological confirmation or advanced imaging data such as positron emission tomography (PET) scan) in which case the principal investigators discretion may determine appropriate timepoint at which study therapy may begin.
* Women of childbearing potential must have a negative beta-human chorionic gonadotropin (HCG) pregnancy test documented within 14 days prior to registration. The effects of Zotiraciclib (TG02) on the developing human fetus are unknown. For this reason, women of childbearing potential must not be pregnant, must not be breast-feeding, and must practice adequate contraception for the duration of the study, and for 30 days after the last dose of study medication.
* Male patients on treatment with Zotiraciclib (TG02) must agree to use an adequate method of contraception for the duration of the study, and for 30 days after the last dose of study medication as the effects of Zotiraciclib (TG02) on the developing human fetus are unknown.
* Patients must agree to enroll on the Neuro-oncology Branch (NOB) Natural History protocol to allow the assessment of molecular tumor markers.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents. However, prior enrollment on a study using investigational agents is acceptable
* Patients with prior bevacizumab use for tumor treatment. Patients who received bevacizumab for symptom management, including but not limited to cerebral edema, pseudoprogression can be included in the study (To date, there have been no effective regimens developed for recurrent malignant gliomas that are refractory to bevacizumab. Inclusion of this patient population may impact the ability to determine the efficacy of Zotiraciclib (TG02) with Temozolomide (TMZ.)
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from providing informed consent.
* Any condition, including the presence of clinically significant laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study. These would include:

  * Active infection (including persistent fever) including known history of human immunodeficiency virus (HIV) or Hepatitis C infection, because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
  * Diseases or conditions that obscure toxicity or dangerously alter drug metabolism
  * Serious concurrent medical illness e.g. symptomatic congestive heart failure
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide and/or Zotiraciclib (TG02).
* Patients with a history of any other cancer (except non-melanoma skin cancer or melanoma in-situ following curative surgical resection; or carcinoma in-situ of the cervix or bladder), unless in complete remission and off all therapy for that disease for a minimum of 3 years, are ineligible.
* Zotiraciclib (TG02) is primarily metabolized by Cytochrome P450 1A2 (CYP1A2) and Cytochrome P450 3A4 (CYP3A4). Patients receiving any medications or substances that are strong inhibitors or inducers of CYP1A2 and/or CYP3A4 are ineligible.
* Patients, who continue to have prolonged corrected QT interval (QTc) (males: greater than 450ms; females: greater than 470ms as calculated by Fridericia s correction formula) despite normal electrolyte balance and discontinuation of medications known to prolong QTc, will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wu, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the Study Protocol, SAP and the Informed Consent Form on ClinicalTrials.gov.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study Protocol, SAP, and Informed Consent Form will be available indefinitely after summary results data is published on clinicaltrials.gov.
Access Criteria: Study Protocol, SAP, and Informed Consent Form will be accessible via clinicaltrials.gov.

REFERENCES:
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0009.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A Phase II study and strategy will be discussed in an upcoming meeting with the FDA to potentially conduct the Phase II as a separate protocol.
Groups:
- ARM 1 Dose Level 0 - (Starting Dose): Temozolomide (TMZ) 125mg/m^2/day, 7 days on and 7 days off; and Zotiraciclib (TG02) 200mg/day on day 1,12,15, 26 per 28-day cycle and one extra dose given 3 days prior to Day 1 cycle 1.
- ARM 1 Dose Level 1 - (Dose Escalation); ARM 1 Dose Level 1 (MTD Level in ARM1): Temozolomide (TMZ) 125mg/m^2/day, 7 days on and 7 days off; and Zotiraciclib (TG02) 250mg/day on day 1,12,15, 26 per 28-day cycle and one extra dose given 3 days prior to Day 1 cycle 1.
- ARM 2 Dose Level 0 (Starting Dose); ARM 2 Dose 0 - (Dose De-escalation): Temozolomide (TMZ) 50mg/m^2 Daily; and Zotiraciclib (TG02) 200mg/day on day 1,12,15, 26 per 28-day cycle and one extra dose given 3 days prior to Day 1 cycle 1.
- ARM 2 Dose 1 - (Dose Escalation); ARM 2 Dose Level I - (Dose De-escalation): Temozolomide (TMZ) 50mg/m^2 Daily; and Zotiraciclib (TG02) 250mg/day on day 1,12,15, 26 per 28-day cycle and one extra dose given 3 days prior to Day 1 cycle 1.
- ARM 2 Dose Level II - (Dose Escalation): Temozolomide (TMZ) 50mg/m^2 Daily; and Zotiraciclib (TG02) 300mg/day on day 1,12,15, 26 per 28-day cycle and one extra dose given 3 days prior to Day 1 cycle 1.
- ARM 2 Dose Level 1 (MTD Level in ARM2): Temozolomide (TMZ) 50mg/m^2 Daily and Zotiraciclib (TG02) 250mg/day on day 1,12,15, 26 per 28-day cycle and one extra dose given 3 days prior to Day 1 cycle 1.
Period: Phase 1 MTD Finding Stage
Arm/Group | ARM 1 Dose Level 0 - (Starting Dose) | ARM 1 Dose Level 1 - (Dose Escalation) | ARM 2 Dose Level 0 (Starting Dose) | ARM 2 Dose 1 - (Dose Escalation) | ARM 2 Dose 0 - (Dose De-escalation) | ARM 2 Dose Level II - (Dose Escalation) | ARM 2 Dose Level I - (Dose De-escalation) | ARM 1 Dose Level 1 (MTD Level in ARM1) | ARM 2 Dose Level 1 (MTD Level in ARM2)
Started | 6 | 13 | 3 | 6 | 3 | 2 | 7 | 0 | 0
Completed | 6 | 12 | 3 | 6 | 3 | 2 | 6 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal of consent | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Phase 1 Cohort Expansion Stage
Arm/Group | ARM 1 Dose Level 0 - (Starting Dose) | ARM 1 Dose Level 1 - (Dose Escalation) | ARM 2 Dose Level 0 (Starting Dose) | ARM 2 Dose 1 - (Dose Escalation) | ARM 2 Dose 0 - (Dose De-escalation) | ARM 2 Dose Level II - (Dose Escalation) | ARM 2 Dose Level I - (Dose De-escalation) | ARM 1 Dose Level 1 (MTD Level in ARM1) | ARM 2 Dose Level 1 (MTD Level in ARM2)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal of consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM 1 Dose Level 0 - (Starting Dose) | ARM 1 Dose Level 1 - (Dose Escalation) | ARM 2 Dose Level 0 (Starting Dose) | ARM 2 Dose 1 - (Dose Escalation) | ARM 2 Dose 0 - (Dose De-escalation) | ARM 2 Dose Level II - (Dose Escalation) | ARM 2 Dose Level I - (Dose De-escalation) | ARM 1 Dose Level 1 (MTD Level in ARM1) | ARM 2 Dose Level 1 (MTD Level in ARM2) | Total
Number analyzed (Participants) | 6 | 13 | 3 | 6 | 3 | 2 | 7 | 6 | 7 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 13 | 3 | 5 | 3 | 2 | 6 | 4 | 5 | 46
  >=65 years | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.47 (18.41) | 48.15 (10.47) | 33.3 (12.93) | 55.2 (14.25) | 38.7 (18.68) | 49.05 (11.1) | 54.46 (9.87) | 56.38 (11.63) | 56.36 (13.15) | 50.38 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 0 | 0 | 1 | 1 | 4 | 0 | 1 | 13
  Male | 4 | 9 | 3 | 6 | 2 | 1 | 3 | 6 | 6 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 4
  Not Hispanic or Latino | 5 | 12 | 3 | 5 | 2 | 2 | 7 | 5 | 7 | 48
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 4
  White | 6 | 12 | 3 | 5 | 1 | 2 | 5 | 4 | 7 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 13 | 3 | 6 | 3 | 2 | 7 | 6 | 7 | 53

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Zotiraciclib in Combination With Dose Dense (dd) Temozolomide (TMZ) in Adult Patients With Recurrent Anaplastic Astrocytoma or Glioblastoma/Gliosarcoma
Description: Maximum tolerated dose of Zotiraciclib (TG02) in combination with dose dense Temozolomide (TMZ) was assessed using the Bayesian Optimal Interval (BOIN) design. The MTD is defined as the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate of 0.35. If there are ties, we select the higher dose level when the isotonic estimate is lower than the target toxicity rate; and we select the lower dose level when the isotonic estimate is greater than the target toxicity rate of 0.35.
Time Frame: 4 weeks after initiation of treatment
Measure: Number; unit: mg/day
Groups:
- All Participants: All participants in ARM 1 in MTD finding stage: Phase (Ph) I Arm 1 Dose Level (DL) 0, and Ph I Arm 1 DL1.
Arm/Group | All Participants
Number analyzed (Participants) | 19
mg/day | 250

2. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Zotiraciclib (TG02) in Combination of Metronomic (mn) Temozolomide (TMZ) in Adult Patients With Recurrent Anaplastic Astrocytoma or Glioblastoma/Gliosarcoma
Description: Maximum tolerated dose of metronomic (mn) Zotiraciclib (TG02) was assessed using the Bayesian Optimal Interval (BOIN) design. The MTD is defined as the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate of 0.35. If there are ties, we select the higher dose level when the isotonic estimate is lower than the target toxicity rate; and we select the lower dose level when the isotonic estimate is greater than the target toxicity rate of 0.35.
Time Frame: 4 weeks after initiation of treatment
Measure: Number; unit: mg/day
Groups:
- All Participants: All participants in ARM2 in MTD finding stage: Phase (Ph) I Arm 2 DL0, Ph I Arm 2 DL1, Ph I Arm 2 Dose 0, Ph I Arm 2 DLII and Ph I DLI.
Arm/Group | All Participants
Number analyzed (Participants) | 21
mg/day | 250

3. Primary Outcome: % of Participants Free of Disease Progression at 4mos Treated w/Zotiraciclib at the Maximum Tolerated Dose in Combination Temozolomide w/Dose Dense Temozolomide Schedules in Adult Patients With Recurrent Anaplastic Astrocytoma or Glioblastoma/Gliosarcoma
Description: We first determined the maximum tolerated dose (MTDs) in each ARM and we then performed the cohort expansion at the MTD in both ARMs separately, until we treated a total of 18 participants at this dose in each ARM. PFS is defined as the duration of time from start of registration to time of progression or death, whichever comes first. Progression was assessed by the Response Assessment in Neuro-Oncology Criteria (RANO). Progression is ≥25% increase in tumor volume compared to baseline in the sum of the products of perpendicular diameters of enhancing lesions compared with the smallest measurement obtained either at baseline or best response with the participant on stable or increasing doses of steroids. Significant increase in T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR) non-enhancing lesions with the participant on stable or increasing doses of steroids (not caused by comorbid events). Any new lesions.
Time Frame: 4 months
Measure: Number; unit: percentage of participants
Groups:
- All Participants: 13 participants in the ARM1 MTD finding stage and 6 participants in the cohort expansion stage: Phase (Ph) I Arm 1 Dose Level (DL) 1
Arm/Group | All Participants
Number analyzed (Participants) | 19
percentage of participants | 40

4. Primary Outcome: % of Participants Free of Disease Progression at 4mos Treated w/Zotiraciclib at the Maximum Tolerated Dose (MTD) in Combination With the Metronomic (mn) Temozolomide (TMZ) in Adult Patients With Recurrent Anaplastic Astrocytoma or Glioblastoma/Gliosarcoma
Description: We first determined the MTDs in each ARM and we then performed the cohort expansion at the MTD in both ARMs separately, until we treated a total of 18 participants at this dose in each ARM. PFS is defined as the duration of time from start of registration to time of progression or death, whichever comes first. Progression was assessed by the Response Assessment in Neuro-Oncology Criteria (RANO). Progression is ≥25% increase in tumor volume compared to baseline in the sum of the products of perpendicular diameters of enhancing lesions compared with the smallest measurement obtained either at baseline or best response with the participant on stable or increasing doses of steroids. Significant increase in T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR) non-enhancing lesions with the participant on stable or increasing doses of steroids (not caused by comorbid events). Any new lesions.
Time Frame: 4 months
Measure: Number; unit: percentage of participants
Groups:
- All Participants: 13 participants in the ARM 2 MTD finding stage and 7 participants in the cohort expansion stage: Phase (Ph) I Arm 2 DL1.
Arm/Group | All Participants
Number analyzed (Participants) | 20
percentage of participants | 25

5. Primary Outcome: Phase II: Progression Free Survival in Subjects Taking Zotiraciclib (TG02) Plus Temozolomide (TMZ) Versus TMZ Alone in Patients With Recurrent World Health Organization (WHO) Grade III or IV Astrocytoma.
Description: Median amount of time subject survives without disease progression after treatment
Time Frame: Disease progression
Population: This outcome measure was not done because a Phase II study and strategy will be discussed in an upcoming meeting with the FDA to potentially conduct the Phase II as a separate protocol.
Groups:
- Phase II: All participants in phase II.
Arm/Group | Phase II
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 15mo(m)/8days(d), 26m, 7m/26d, 13m/17d, 11m/30d, 12m/6d, 19m/11d, 9m/28d and 18m/21d for Group 1-9 respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 Dose Level 0 - (Starting Dose) | ARM 1 Dose Level 1 - (Dose Escalation) | ARM 2 Dose Level 0 (Starting Dose) | ARM 2 Dose 1 - (Dose Escalation) | ARM 2 Dose 0 - (Dose De-escalation) | ARM 2 Dose Level II - (Dose Escalation) | ARM 2 Dose Level I - (Dose De-escalation) | ARM 1 Dose Level 1 (MTD Level in ARM1) | ARM 2 Dose Level 1 (MTD Level in ARM2)
Number analyzed (Participants) | 6 | 13 | 3 | 6 | 3 | 2 | 7 | 6 | 7
Participants | 6 | 13 | 3 | 6 | 3 | 2 | 7 | 6 | 7

7. Other Pre Specified Outcome: Phase I: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: DLT is defined as any adverse events attributed to the study drug. For example, Grade 4 neutropenia lasting 5 days or more. Febrile neutropenia defined as grade 3-4 neutropenia with fever ≥38.5ºC and/or infection requiring antibiotic or antifungal treatment. Nausea or vomiting that responds to symptomatic therapy and lasts ≤7 days. Fatigue that responds to symptomatic therapy and lasts ≤7 days. And weight gain (in patients on steroids).
Time Frame: 4 weeks after initiation of treatment
Population: Arm2 DI: After prot. amend. previously defined gr 4 lymphopenia was no longer counted as DLT. 2/3 DLTs listed here are no longer DLTs. Arm2 D0:Prot. amend occurred after this dose de-escal. Re-eval. of DLT rate at DL1 led to the next dose escal. Analysis not applic. for Arm1 DL1& Arm2D. Arm1 DL1:Per study design, pts in expans. stage are not analyzed for DLT. Arm2 DL1:Per study design, pts in expans. stage are not analyzed for DLT;as part of the expans. no pt in this grp were analyzed for DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1 Dose Level 0 - (Starting Dose) | ARM 1 Dose Level 1 - (Dose Escalation) | ARM 2 Dose Level 0 (Starting Dose) | ARM 2 Dose 1 - (Dose Escalation) | ARM 2 Dose 0 - (Dose De-escalation) | ARM 2 Dose Level II - (Dose Escalation) | ARM 2 Dose Level I - (Dose De-escalation) | ARM 1 Dose Level 1 (MTD Level in ARM1) | ARM 2 Dose Level 1 (MTD Level in ARM2)
Number analyzed (Participants) | 6 | 13 | 3 | 6 | 3 | 2 | 7 | 0 | 0
Participants | 1 | 3 | 0 | 3 | 1 | 1 | 4 |  |

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 15mo(m)/8days(d), 26m, 7m/26d, 13m/17d, 11m/30d, 12m/6d, 19m/11d, 9m/28d and 18m/21d for Group 1-9 respectively.
Groups:
- ARM 1 Dose Level 0 (Starting Dose): Temozolomide (TMZ) 125mg/m^2/day, 7 days on and 7 days off; and Zotiraciclib (TG02) 200mg/day on day 1,12,15, 26 per 28-day cycle and one extra dose given 3 days prior to Day 1 cycle 1.
- ARM 1 Dose Level 1 (Dose Escalation); ARM 1 Dose Level 1 (MTD Level in ARM1): Temozolomide (TMZ) 125mg/m^2/day, 7 days on and 7 days off; and Zotiraciclib (TG02) 250mg/day on day 1,12,15, 26 per 28-day cycle and one extra dose given 3 days prior to Day 1 cycle 1.
- ARM 2 Dose 1 (Dose Escalation); ARM 2 Dose Level I (Dose De-escalation): Temozolomide (TMZ) 50mg/m^2 Daily; and Zotiraciclib (TG02) 250mg/day on day 1,12,15, 26 per 28-day cycle and one extra dose given 3 days prior to Day 1 cycle 1.
- ARM 2 Dose 0 (Dose De-escalation): Temozolomide (TMZ) 50mg/m^2 Daily; and Zotiraciclib (TG02) 200mg/day on day 1,12,15, 26 per 28-day cycle and one extra dose given 3 days prior to Day 1 cycle 1.
- ARM 2 Dose Level II (Dose Escalation): Temozolomide (TMZ) 50mg/m^2 Daily; and Zotiraciclib (TG02) 300mg/day on day 1,12,15, 26 per 28-day cycle and one extra dose given 3 days prior to Day 1 cycle 1.
Arm/Group | ARM 1 Dose Level 0 (Starting Dose) | ARM 1 Dose Level 1 (Dose Escalation) | ARM 2 Dose Level 0 (Starting Dose) | ARM 2 Dose 1 (Dose Escalation) | ARM 2 Dose 0 (Dose De-escalation) | ARM 2 Dose Level II (Dose Escalation) | ARM 2 Dose Level I (Dose De-escalation) | ARM 1 Dose Level 1 (MTD Level in ARM1) | ARM 2 Dose Level 1 (MTD Level in ARM2)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/13 | 2/3 | 0/6 | 1/3 | 0/2 | 1/7 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/6 | 8/13 | 1/3 | 4/6 | 1/3 | 2/2 | 2/7 | 2/6 | 2/7
Other Adverse Events (participants affected / at risk) | 6/6 | 13/13 | 3/3 | 6/6 | 3/3 | 2/2 | 7/7 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 1 Dose Level 0 (Starting Dose) (N=6) | ARM 1 Dose Level 1 (Dose Escalation) (N=13) | ARM 2 Dose Level 0 (Starting Dose) (N=3) | ARM 2 Dose 1 (Dose Escalation) (N=6) | ARM 2 Dose 0 (Dose De-escalation) (N=3) | ARM 2 Dose Level II (Dose Escalation) (N=2) | ARM 2 Dose Level I (Dose De-escalation) (N=7) | ARM 1 Dose Level 1 (MTD Level in ARM1) (N=6) | ARM 2 Dose Level 1 (MTD Level in ARM2) (N=7)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema cerebral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, Planned surgical procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 1 Dose Level 0 (Starting Dose) (N=6) | ARM 1 Dose Level 1 (Dose Escalation) (N=13) | ARM 2 Dose Level 0 (Starting Dose) (N=3) | ARM 2 Dose 1 (Dose Escalation) (N=6) | ARM 2 Dose 0 (Dose De-escalation) (N=3) | ARM 2 Dose Level II (Dose Escalation) (N=2) | ARM 2 Dose Level I (Dose De-escalation) (N=7) | ARM 1 Dose Level 1 (MTD Level in ARM1) (N=6) | ARM 2 Dose Level 1 (MTD Level in ARM2) (N=7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (18) | 11 (29) | 1 (13) | 6 (14) | 2 (3) | 1 (1) | 3 (10) | 4 (9) | 6 (14)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (5) | 5 (6) | 2 (5) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (11) | 8 (13) | 1 (3) | 4 (6) | 1 (2) | 2 (2) | 3 (5) | 2 (3) | 5 (7)
Ataxia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 1 (2) | 1 (3) | 2 (2) | 1 (2) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (5) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (3) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (24) | 9 (28) | 3 (5) | 2 (16) | 1 (1) | 1 (1) | 4 (13) | 2 (4) | 6 (12)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Facial muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (7) | 1 (2) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 3 (6) | 4 (4) | 3 (6)
Fatigue (General disorders) | 4 (8) | 7 (15) | 3 (3) | 5 (11) | 1 (1) | 1 (1) | 5 (14) | 3 (5) | 5 (8)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (6) | 6 (7) | 2 (2) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 3 (3)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 5 (8) | 1 (3) | 4 (9) | 0 (0) | 1 (1) | 4 (13) | 1 (1) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (30) | 9 (34) | 3 (21) | 6 (31) | 0 (0) | 2 (13) | 5 (22) | 6 (28) | 7 (44)
Malaise (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (12) | 7 (12) | 2 (8) | 4 (7) | 3 (8) | 1 (1) | 5 (8) | 1 (1) | 6 (9)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (23) | 7 (38) | 2 (17) | 3 (11) | 1 (11) | 1 (5) | 4 (20) | 5 (17) | 7 (37)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Platelet count decreased (Investigations) | 4 (6) | 10 (12) | 0 (0) | 6 (10) | 1 (5) | 1 (8) | 2 (6) | 4 (10) | 4 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (3) | 2 (3)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (10) | 3 (12) | 1 (6) | 4 (8) | 1 (1) | 2 (3) | 5 (12) | 1 (1) | 3 (6)
Weight gain (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 5 (32) | 12 (48) | 3 (21) | 6 (18) | 1 (8) | 2 (15) | 5 (31) | 6 (21) | 7 (57)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT02942264/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT02942264/ICF_001.pdf